CLINICAL TRIAL: NCT02262871
Title: Randomized Cross-over Physiologic Study of High Flow Nasal Oxygen Cannula Versus Non-invasive Ventilation in Cystic Fibrosis. The HIFEN Study
Brief Title: HFN Versus NIV in Cystic Fibrosis. The HIFEN Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB14-338
Record Dates: First submitted 2014-10-07; First posted 2014-10-13 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; High-flow nasal oxygen cannula; Non-invasive ventilation; Respiratory distress; Oxygen therapy
MeSH Terms: conditions — Cystic Fibrosis; Dyspnea | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CF patients HFN (Experimental): CF patients who meet the eligibility criteria will be randomized to receive HFN and then crossover to other device.
  Interventions: Device: High flow nasal oxygen cannula
- CF patients NIV (Experimental): CF patients who meet the eligibility criteria will be randomized to receive NIV and then crossover to other device.
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: High flow nasal oxygen cannula — HFN will be set with an inspiratory flow rate at 45-55 L/min (maximal tolerated flow), temperature at 37°C or 34°C if perceived as too warm, and fraction on inspired oxygen (FiO2) will be adjusted to achieve an oxygen saturation (SpO2) of at least 92%.
  Arms: CF patients HFN
Device: Noninvasive ventilation — The setting of NIV will be appropriately adjusted, based on the clinical assessment of the respiratory therapist in charge and will not be modified during the test.
  Arms: CF patients NIV

SUMMARY:
Many patients with cystic fibrosis (CF) require hospitalization and/or Intensive Care Unit (ICU) admission because of acute exacerbation of chronic respiratory failure or for any acute deterioration of clinical status. Non-invasive ventilation (NIV) is the first option for the clinical management of CF patients with moderate-to-severe respiratory distress and NIV has been shown to improve gas exchange, reduce respiratory muscle work and improve pulmonary function in patients with obstructive lung disease in general and those with acute CF exacerbation. High-flow nasal oxygen cannula (HFN) is a relatively new system providing heated and humidified, high-flow (50L/min) oxygen through the nostrils. This device provides a small positive pressure, probably washes-out the pharyngeal dead space, reduces inspiratory resistance, and possibly facilitates secretion clearance. The technique is very well tolerated. From a physiologic standpoint, this device could help CF patients by improving gas exchange, reducing respiratory workload, and facilitating mucus clearance. Non-interrupted delivery may be possible given better clinical tolerance in contrast with bi-level positive pressure NIV. Whether the short-term physiological efficacy of HFN is comparable to NIV is unknown and there is no study on the benefit of HFN in CF patients.

The aim of this study is to compare the physiological effects of HFN and NIV in CF patients requiring ventilatory support. Our hypothesis is that HFN will not be inferior to NIV, as evaluated by breathing pattern, gas exchange, and respiratory workload and will decrease dead space. In addition, comfort and preference between the two techniques will be evaluated.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Cystic fibrosis as defined by clinical features in conjunction with 2 CF causing mutations and/or 2 sweat tests with sweat chloride > 60 mmol/l
* Clinical indication for NIV based on at least one of the following criteria:

  * Signs of clinical respiratory distress - RR > 24/min, accessory muscle use, or increased dyspnea
  * Progressive increase in arterial PCO2
  * Nocturnal hypoventilation treated by NIV but requiring daytime NIV because of clinical worsening

Exclusion criteria:

* Active massive hemoptysis
* Pneumothorax with pleural drainage and persistent air leak
* Hemodynamic instability requiring vasopressors
* Uncooperative
* Recent upper airway or esophageal surgery
* Patients with skin or chest wall or abdominal trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
The decrease of diaphragmatic workload (thickening fraction of the diaphragm) | 30 minutes

SECONDARY OUTCOMES:
Respiratory parameters | 30 minutes
  respiratory rate (RR), minute ventilation
Gas exchange | 30 minutes
  pulse oximetry, transcutaneous carbon dioxide partial pressure (PCO2)
Electromyographic activity of the diaphragm | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, Dr., Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Result] Davies JC, Alton EW, Bush A. Cystic fibrosis. BMJ. 2007 Dec 15;335(7632):1255-9. doi: 10.1136/bmj.39391.713229.AD. No abstract available. PMID 18079549
- [Result] Pittman JE, Cutting G, Davis SD, Ferkol T, Boucher R. Cystic fibrosis: NHLBI Workshop on the Primary Prevention of Chronic Lung Diseases. Ann Am Thorac Soc. 2014 Apr;11 Suppl 3(Suppl 3):S161-8. doi: 10.1513/AnnalsATS.201312-444LD. PMID 24754825
- [Result] Flume PA. Pulmonary complications of cystic fibrosis. Respir Care. 2009 May;54(5):618-27. doi: 10.4187/aarc0443. PMID 19393106
- [Result] Nick JA, Chacon CS, Brayshaw SJ, Jones MC, Barboa CM, St Clair CG, Young RL, Nichols DP, Janssen JS, Huitt GA, Iseman MD, Daley CL, Taylor-Cousar JL, Accurso FJ, Saavedra MT, Sontag MK. Effects of gender and age at diagnosis on disease progression in long-term survivors of cystic fibrosis. Am J Respir Crit Care Med. 2010 Sep 1;182(5):614-26. doi: 10.1164/rccm.201001-0092OC. Epub 2010 May 6. PMID 20448091
- [Result] Belkin RA, Henig NR, Singer LG, Chaparro C, Rubenstein RC, Xie SX, Yee JY, Kotloff RM, Lipson DA, Bunin GR. Risk factors for death of patients with cystic fibrosis awaiting lung transplantation. Am J Respir Crit Care Med. 2006 Mar 15;173(6):659-66. doi: 10.1164/rccm.200410-1369OC. Epub 2005 Dec 30. PMID 16387803
- [Result] Sood N, Paradowski LJ, Yankaskas JR. Outcomes of intensive care unit care in adults with cystic fibrosis. Am J Respir Crit Care Med. 2001 Feb;163(2):335-8. doi: 10.1164/ajrccm.163.2.2003076. PMID 11179102
- [Result] Jones A, Bilton D, Evans TW, Finney SJ. Predictors of outcome in patients with cystic fibrosis requiring endotracheal intubation. Respirology. 2013 May;18(4):630-6. doi: 10.1111/resp.12051. PMID 23323684
- [Result] Fauroux B, Burgel PR, Boelle PY, Cracowski C, Murris-Espin M, Nove-Josserand R, Stremler N, Derlich L, Giovanetti P, Clement A; Chronic Respiratory Insufficiency Group of the French National Cystic Fibrosis Federation. Practice of noninvasive ventilation for cystic fibrosis: a nationwide survey in France. Respir Care. 2008 Nov;53(11):1482-9. PMID 18957151
- [Result] Fauroux B. Why, when and how to propose noninvasive ventilation in cystic fibrosis? Minerva Anestesiol. 2011 Nov;77(11):1108-14. Epub 2011 May 20. PMID 21602746
- [Result] Madden BP, Kariyawasam H, Siddiqi AJ, Machin A, Pryor JA, Hodson ME. Noninvasive ventilation in cystic fibrosis patients with acute or chronic respiratory failure. Eur Respir J. 2002 Feb;19(2):310-3. doi: 10.1183/09031936.02.00218502. PMID 11866011
- [Result] Fauroux B, Nicot F, Essouri S, Hart N, Clement A, Polkey MI, Lofaso F. Setting of noninvasive pressure support in young patients with cystic fibrosis. Eur Respir J. 2004 Oct;24(4):624-30. doi: 10.1183/09031936.04.0000137603. PMID 15459142
- [Result] Granton JT, Kesten S. The acute effects of nasal positive pressure ventilation in patients with advanced cystic fibrosis. Chest. 1998 Apr;113(4):1013-8. doi: 10.1378/chest.113.4.1013. PMID 9554640
- [Result] Serra A, Polese G, Braggion C, Rossi A. Non-invasive proportional assist and pressure support ventilation in patients with cystic fibrosis and chronic respiratory failure. Thorax. 2002 Jan;57(1):50-4. doi: 10.1136/thorax.57.1.50. PMID 11809990
- [Result] Young AC, Wilson JW, Kotsimbos TC, Naughton MT. Randomised placebo controlled trial of non-invasive ventilation for hypercapnia in cystic fibrosis. Thorax. 2008 Jan;63(1):72-7. doi: 10.1136/thx.2007.082602. Epub 2007 Aug 3. PMID 17675317
- [Result] Ricard JD. High flow nasal oxygen in acute respiratory failure. Minerva Anestesiol. 2012 Jul;78(7):836-41. Epub 2012 Apr 24. PMID 22531566
- [Result] Cuquemelle E, Pham T, Papon JF, Louis B, Danin PE, Brochard L. Heated and humidified high-flow oxygen therapy reduces discomfort during hypoxemic respiratory failure. Respir Care. 2012 Oct;57(10):1571-7. doi: 10.4187/respcare.01681. Epub 2012 Mar 12. PMID 22417569
- [Result] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Result] Rittayamai N, Tscheikuna J, Rujiwit P. High-flow nasal cannula versus conventional oxygen therapy after endotracheal extubation: a randomized crossover physiologic study. Respir Care. 2014 Apr;59(4):485-90. doi: 10.4187/respcare.02397. Epub 2013 Sep 17. PMID 24046462
- [Result] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Result] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Result] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Result] Vignaux L, Vargas F, Roeseler J, Tassaux D, Thille AW, Kossowsky MP, Brochard L, Jolliet P. Patient-ventilator asynchrony during non-invasive ventilation for acute respiratory failure: a multicenter study. Intensive Care Med. 2009 May;35(5):840-6. doi: 10.1007/s00134-009-1416-5. Epub 2009 Jan 29. PMID 19183949
- [Derived] Sklar MC, Dres M, Rittayamai N, West B, Grieco DL, Telias I, Junhasavasdikul D, Rauseo M, Pham T, Madotto F, Campbell C, Tullis E, Brochard L. High-flow nasal oxygen versus noninvasive ventilation in adult patients with cystic fibrosis: a randomized crossover physiological study. Ann Intensive Care. 2018 Sep 5;8(1):85. doi: 10.1186/s13613-018-0432-4. PMID 30187270